CLINICAL TRIAL: NCT01505413
Title: Phase 2 Study of GEMOX-T in Previously Untreated Patients With Advanced Pancreatic Cancer
Brief Title: Phase 2 Study of Erlotinib, Gemcitabine and Oxaliplatin Combination Chemotherapy to Advanced Pancreatic Cancer
Acronym: GEMOX-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jina Yun, Division of Oncology-Hematology Department of Internal medicine, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yun-11349
Record Dates: First submitted 2012-01-02; First posted 2012-01-06 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer
Keywords: advanced unresectable or metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tarceva, Gemcitabine, Oxaliplatin (Experimental): * Erlotinib 100 mg po qd daily AND
  * Gemcitabine 1000 mg/m² with 150mL of normal saline intravenously infusion over 100min on Day 1
  * Oxaliplatin 100 mg/m2 with 500mL of 5DW intravenously a 2-hour infusion on D2 Every 2 weeks
  Each two weeks is a cycle. If at end of 12 cycles response continues, will administer Gemcitabine and erlotinib until progression.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 100 mg po qd daily
  Other Names: tarceva
Drug: Gemcitabine — Gemcitabine 1000 mg/m² with 150mL of normal saline intravenously infusion over 100min on Day 1
  Other Names: gemza; gemcibine
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 with 500mL of 5DW intravenously a 2-hour infusion on D2
  Other Names: oxalitin

SUMMARY:
Erlotinib is an orally available, reversible tyrosine kinase inhibitor of epidermal growth factor receptor (EGFR). Association of chemoresistance with the activity of certain tyrosine kinases (e.g. ErbB-1 and Src) has been described for pancreatic cancer and makes a strong case for combining gemcitabine with tyrosine kinase inhibitors. In a phase III trial, the addition of erlotinib to gemcitabine improved survival compared with gemcitabine alone in advanced pancreatic cancer (MJ Moor et al). Also, gemcitabine in combination with oxaliplatin is superior to gemcitabine alone in terms of progression free survival and response rate in one phase III trial (Louvet et al). Taken together, combining erlotinib with gemcitabine and oxaliplatin may further improve the overall survival and clinical benefit of advanced pancreatic cancer.

DETAILED DESCRIPTION:
Open, uncontrolled, multicenter, phase II study

This study will enroll previous chemo-naïve patients with locally advanced unresectable or metastatic pancreatic cancer.

Study regimen:

* Erlotinib 100 mg po qd daily AND
* Gemcitabine 1000 mg/m² with 150mL of normal saline intravenously infusion over 100min on Day 1
* Oxaliplatin 100 mg/m2 with 500mL of 5DW intravenously a 2-hour infusion on D2 Every 2 weeks

Each two weeks is a cycle. If at end of 12 cycles response continues, will administer Gemcitabine and erlotinib until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. ECOG performance status of ≤2
3. Histologically confirmed adenocarcinoma of the pancreas
4. The disease is Locally advanced deemed by the surgeon to be unresectable, or metastatic disease.
5. Prior chemotherapy is not permitted, except for fluorouracil given concurrently as a radiosensitizer.
6. Patients must have normal organ function evidenced by

   * Number of absolute neutrophil counts (ANC) > 1.5 x 109/L
   * Number of thrombocytes > 100 x 109/L
   * Total bilirubin < 1.5 x upper limit of normal (although patients with a Total bilirubin count between 1.5 and 3 x upper limit of normal in whom a decrease is anticipated, ex. Biliary stent insertion)ALAT, ASAT < 3 x upper limit of normal (in case of liver metastasis, 5 x upper limit of normal)
   * Alkaline phosphatase < 3 x upper limit of normal (in case of liver metastasis, 5 x upper limit of normal)
7. Pain should be controlled for at least two weeks without an increase in the narcotic consumption.
8. Biliary obstruction should be controlled for at least two weeks evident by stable or improving liver function tests especially total bilirubin.
9. Patient has signed a Patient Informed Consent Form.
10. For all females of childbearing potential, a negative pregnancy test must be obtained within 72 hours before starting therapy.
11. Is able to take medications orally
12. A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in spiral CT or multidetector CT (MD CT) or 20 mm or longer in conventional CT (it should be used by a consistent method during the study period)

Exclusion Criteria:

1. Tumor type other than adenocarcinoma
2. Evidence of uncontrolled CNS disease (patients with controlled CNS disease for 4 weeks using the same imaging method and for whom are off steroid will be eligible)
3. Uncontrolled Nausea and Vomiting
4. Diagnosis of other malignancy in the last 5 years excluding non-melanoma skin cancer and in -situ cervical cancer.
5. Subjects unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow- up visits and unlikelihood of completing the study.
6. Any known history of hypersensitivity to the study drugs.
7. Pregnant or lactating women.
8. Symptomatic peripheral sensory neuropathy (NCI CTCAE v3.0 ≥ grade 2)
9. Other serious illness or medical condition, notably heart or lung failure, active uncontrolled infection
10. Prior radiotherapy was administered to target lesions selected for this study, or radiotherapy to the non-target lesions has been completed within 4 weeks before being included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response rate | 24 months (01/2011 and end of study 01/2013)
  Responses are assessed every 2 cycles according to RECIST; the imaging tests are performed in a week preceding the corresponding cycles, and can also be repeated at any other time if clinically indicated, for example, to confirm disease progression. At any time, patients with progressive disease are withdrawn.

SECONDARY OUTCOMES:
disease control rate(SD,PR,CR) | 24 months (01/2011 and end of study 01/2013)
  Responses are assessed every 2 cycles according to RECIST; the imaging tests are performed in a week preceding the corresponding cycles, and can also be repeated at any other time if clinically indicated, for example, to confirm disease progression. At any time, patients with progressive disease are withdrawn.
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Taek Lee, Dr, Study Director — Soonchunhyang University Hospital; Hee Sook Park, Dr, Study Director — Soonchunhyang University Hospital; Dae Sik Hong, Dr, Study Director — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea